CLINICAL TRIAL: NCT04527991
Title: A Randomized Open-Label Phase III Study of Sacituzumab Govitecan Versus Treatment of Physician's Choice in Subjects With Metastatic or Locally Advanced Unresectable Urothelial Cancer
Brief Title: Study of Sacituzumab Govitecan Versus Physician's Choice of Treatment in Participants With Urothelial Cancer That Cannot Be Removed or Has Spread
Acronym: TROPiCS-04
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMMU-132-13; 2024-513870-23 (Other: EU CT Number)
Record Dates: First submitted 2020-08-19; First posted 2020-08-27 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced or Metastatic Unresectable Urothelial Cancer
MeSH Terms: interventions — sacituzumab govitecan; Paclitaxel; Docetaxel; vinflunine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sacituzumab Govitecan-hziy (Experimental): Participants will receive 10 mg/kg of sacituzumab govitecan-hziy intravenously on Day 1 and Day 8 of 21-day cycles.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Treatment of Physician's Choice (Active Comparator): Participants will have the choice of receiving paclitaxel, docetaxel, or vinflunine at standard of care (SOC) doses of 175, 75, and 320 mg/m^2 respectively, every 3 weeks on Day 1 of 21-day cycles.
  Interventions: Drug: Paclitaxel; Drug: Docetaxel; Drug: Vinflunine

INTERVENTIONS:
Drug: Sacituzumab Govitecan-hziy — Administered intravenously
  Other Names: IMMU-132; Trodelvy™; GS-0132
  Arms: Sacituzumab Govitecan-hziy
Drug: Paclitaxel — Administered intravenously
  Other Names: Taxol®
  Arms: Treatment of Physician's Choice
Drug: Docetaxel — Administered intravenously
  Other Names: Taxotere®
  Arms: Treatment of Physician's Choice
Drug: Vinflunine — Administered intravenously
  Other Names: Javlor ®
  Arms: Treatment of Physician's Choice

SUMMARY:
The primary objective of this study is to assess overall survival (OS) with sacituzumab govitecan-hziy in comparison with treatment of physician's choice (TPC) in participants with metastatic or locally advanced unresectable urothelial cancer (UC).

ELIGIBILITY:
Key Inclusion Criteria:

1. Individuals with histologically documented metastatic or locally advanced unresectable UC defined as

   * Tumor (T) 4b, any node (N) or
   * Any T, N 2-3 Tumors of upper and lower urinary tract are permitted. Mixed histologic types are allowed if urothelial is the predominant histology.
2. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1.
3. Individuals with progression or recurrence following receipt of platinum-containing regimen and anti programmed cell death protein 1/programmed death-ligand 1 (PD-1/PD-L1) therapy for metastatic or locally advanced unresectable disease will be enrolled.

   * a. Individuals with recurrence or progression ≤12 months following completion of cisplatin-containing chemotherapy given in the neo-adjuvant/adjuvant setting may utilize that line of therapy to be eligible for the study. The 12-month period is counted from completion of surgical intervention or platinum therapy, respectively. These individuals must receive anti PD-1/PD-L1 therapy in the metastatic or locally advanced unresectable setting to be eligible.
   * b. Individuals who received either carboplatin or anti PD-1/PD-L1 therapy in the neo- adjuvant/adjuvant setting will not be able to count that line of therapy towards eligibility for the study.
   * c. Cisplatin ineligible individuals who meet one of the below criteria and who were treated with carboplatin in the metastatic or locally advanced unresectable settings may count that line of therapy towards eligibility. They must then have received anti PD-1/PD-L1 therapy in metastatic or locally advanced unresectable setting to be eligible for the study.

     * Cisplatin ineligibility is defined as meeting one of the following criteria:

       * 1. Creatinine Clearance < 60 mL/min
       * 2. Grade ≥ 2 Audiometric Hearing Loss
       * 3. Grade ≥ 2 Peripheral Neuropathy
       * 4. New York Heart Association (NYHA) Class III heart failure
       * 5. ECOG PS ≥ 2
   * d. Anti PD-1/PD-L1 therapy administered as part of maintenance therapy may be counted towards eligibility for the study
   * e. Individuals who have progressed after receiving enfortumab vedotin in prior lines of therapy, and individuals who are either ineligible or unable to tolerate enfortumab vedotin therapy, are eligible to enroll in the study
   * f. Individuals who received only concurrent chemoradiation for bladder preservation without further systemic therapy are not eligible to enroll in the study. The substitution of carboplatin for cisplatin does not constitute a new regimen provided no new chemotherapeutic agents were added to the regimen and no progression was noted prior to the change in platinum.
4. Individuals with previously treated brain metastases may participate in the study provided they have stable CNS disease for at least 4 weeks prior to the first dose of study drug and stabilization of all neurologic symptoms, have no evidence of new or enlarging brain metastases, and are not using steroids >20 mg of prednisone (or equivalent) daily for brain metastases for at least 7 days prior to first dose of the study drug.
5. Adequate hematologic counts without transfusion or growth factor support within 2 weeks of study drug initiation (hemoglobin ≥ 9 g/dL, absolute neutrophil count (ANC) ≥1,500/mm^3, and platelets ≥100,000/µL).
6. Adequate hepatic function (bilirubin ≤1.5x institutional upper limit of normal (IULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x IULN or ≤ 5 x IULN if known liver metastases and serum albumin >3 g/dL).

   Docetaxel will only be option in TPC arm for Individuals with a total bilirubin ≤1 x IULN, and an AST and/or ALT ≤1.5x IULN if alkaline phosphatase is also >2.5 x IULN.
7. Creatinine clearance ≥30 mL/min as assessed by the Cockcroft-Gault equation or other validated instruments (e.g. Modification of Diet in Renal Disease (MDRD) equation).
8. Females of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study drug. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Females of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 6 months after the last dose of study drug. Individuals of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >2 years.
10. Males must agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study therapy.

Key Exclusion Criteria:

1. Females who are pregnant or lactating.
2. Have had a prior anti-cancer monoclonal antibody (mAb)/ antibody-drug conjugate (ADC) within 4 weeks prior to Cycle 1 Day 1 (C1D1) or have had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to C1D1. Individuals participating in observational studies are eligible.
3. Have received prior chemotherapy for UC with any available SOC therapies in the control arm (i.e., both prior paclitaxel and docetaxel in regions where vinflunine is not an approved therapy, or prior paclitaxel, docetaxel and vinflunine in regions where vinflunine is approved and is commercially available).
4. Have not recovered (i.e., ≤ Grade 1) from AEs due to previously administered chemotherapeutic agent.

   * Note: Individuals with ≤ Grade 2 neuropathy or any grade of alopecia are an exception to this criterion and will qualify for the study.
   * Note: If Individuals received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study therapy.
5. Have previously received topoisomerase 1 inhibitors.
6. Have an active second malignancy.

   • Note: Individuals with a history of malignancy that have been completely treated and with no evidence of active cancer for 3 years prior to enrollment, or individuals with surgically cured tumors with low risk of recurrence are allowed to enroll in the study after discussion with the medical monitor.
7. Have active cardiac disease, defined as:

   * Myocardial infarction or unstable angina pectoris within 6 months of C1D1.
   * History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication); history of QT interval prolongation.
   * NYHA Class III or greater congestive heart failure or left ventricular ejection fraction of <40%.
8. Have active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or gastrointestinal (GI) perforation within 6 months of enrollment.
9. Have an active serious infection requiring anti-infective therapy (Contact medical monitor for clarification).
10. Have known history of Human Immunodeficiency Virus (HIV)-1/2 with undetectable viral load and on medications that may interfere with SN-38 metabolism.
11. Have active Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV). In individuals with a history of HBV or HCV, individuals with a detectable viral load will be excluded.
12. Have other concurrent medical or psychiatric conditions that, in the investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
13. Have inability to tolerate or are allergic to any potential TPC agent or sacituzumab govitecan-hziy or unable or unwilling to receive the doses specified in the protocol.
14. Have inability to complete all specified study procedures for any reason.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 3.5 years
  OS is defined as time from the date of randomization to the date of death, regardless of cause.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) by Investigator Assessment | Up to 3.5 years
  PFS is defined as the time from the date of randomization to the date of the first objectively documented disease progression, per response evaluation criteria in solid tumors version 1.1 (RECIST v1.1) criteria, as determined by investigator assessment, or death regardless of cause, whichever occurs first.
Progression-Free Survival (PFS) by Blinded Independent Central Review (BICR) | Up to 3.5 years
  PFS is defined as the time from the date of randomization to the date of the first objectively documented disease progression, per RECIST v1.1 criteria as determined by BICR, or death regardless of cause, whichever occurs first.
Objective Response Rate (ORR) by Investigator Assessment | Up to 3.5 years
  ORR is defined as the proportion of participants who achieved a complete response or partial response as best overall response (BOR). BOR is determined per RECIST 1.1 as determined by investigator assessment.
Objective Response Rate (ORR) by BICR | Up to 3.5 years
  ORR is defined as the proportion of participants who achieved a complete response or partial response as best overall response (BOR). BOR is determined per RECIST 1.1 as determined by BICR.
Clinical Benefit Rate (CBR) by Investigator Assessment | Up to 3.5 years
  CBR is defined as the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease for greater than or equal to 6 months to therapeutic intervention in a clinical study. CBR will be determined per RECIST v1.1 by investigator assessment.
Clinical Benefit Rate (CBR) by BICR | Up to 3.5 years
  CBR is defined as the percentage of participants with advanced or metastatic cancer who have achieved complete response, partial response and stable disease for greater than or equal to 6 months to therapeutic intervention in a clinical study. CBR will be determined per RECIST v1.1 by BICR.
Duration of Objective Tumor Response (DOR) by Investigator Assessment | Up to 3.5 years
  DOR is defined as the time from the date when the criteria is first met for a complete response or partial response to the first date that disease progression is documented per RECIST 1.1 as determined by investigator assessment, or date of death, whichever occurs first.
Duration of Objective Tumor Response (DOR) by BICR | Up to 3.5 years
  DOR is defined as the time from the date when the criteria is first met for a complete response or partial response to the first date that disease progression is documented per RECIST 1.1 as determined by BICR, or date of death, whichever occurs first.
Percentage of Participants Experiencing any Treatment Emergent Adverse Events | Up to 3.5 years
Percentage of Participants Experiencing any Serious Treatment Emergent Adverse Events | Up to 3.5 years
Percentage of Participants Experiencing any Clinically Significant Laboratory Abnormalities | Up to 3.5 years
European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30) Score | Up to 3.5 years
  The EORTC QLQ-C30 is a questionnaire to assess quality of life of cancer patients, it is composed of 30 questions (items) resulting in 5 functional scales, 1 global health status scale, 3 symptom scales, and 6 single items. Scoring of the QLQ-C30 is performed according to QLQ-C30 Scoring manual. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the participant), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the participant).
European Quality of Life 5-Dimensions 5 Levels Instrument (EuroQOL EQ-5D-5L) Score | Up to 3.5 years
  The EQ-5D-5L is a standard measure of health-related quality of life. The tool consists of the EQ-5D-5L descriptive part and the EQ visual analogue scale (VAS). The descriptive part comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each of these 5 dimensions has 5 levels (no problem, slight problems, moderate problems, severe problems, and extreme problems). Results for each of the 5 dimensions are combined into a 5-digit number to describe the participant's health state.
  The EQ-VAS records the participant's health on a 0-100 mm VAS scale, with 0 indicating "the worst health you can imagine" and 100 indicating "the best health you can imagine." Higher scores of EQ VAS indicate better health.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (234):
- United States (21):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - UCLA Hematology/ Oncology, Los Angeles, California
  - University of California Irvine (UCIMC), Orange, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Boca Raton Clinical Research Global USA - Plantation, Plantation, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medical College, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oklahoma Cancer Specialists and Research Institute (OCSRI), Tulsa, Oklahoma
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - Thompson Oncology Group - Knoxville Downtown, Knoxville, Tennessee
  - University Cancer Specialists - Knoxville, Knoxville, Tennessee
  - Harold C. Simmons Comprehensive Cancer Center, Dallas, Texas
  - Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Seattle Cancer Care Alliance (SCCA), Seattle, Washington
  - Summit Cancer Centers, Spokane, Washington
- Australia (13):
  - Chris O'Brien Lifehouse, North Ryde, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Icon Cancer Centre Wesley, Auchenflower, Queensland
  - Southern Adelaide Local Health Network Incorporated, Bedford Park, South Australia
  - Ashford Cancer Centre Research - ICON Cancer Centre Adelaide, Kurralta Park, South Australia
  - ICON Cancer Centre Hobart, Hobart, Tasmania
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sunshine Hospital, Saint Albans, Victoria
  - Liverpool Hospital, Nedlands, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Austria (3):
  - Universitätsklinik für Innere Medizin Graz, Graz
  - Ordensklinikum Linz GmbH Barmherzige Schwestern, Linz
  - Krankenhaus Der Barmherzigen Bruder Wien, Vienna
- Belgium (5):
  - Grand Hôpital De Charleroi - Notre Dame, Charleroi
  - Az Maria Middelares Ghent, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Bulgaria (2):
  - Multiprofile Hospital for Active Treatment Heart and Brain EAD, Pleven
  - Specialized Hospital for Active Treatment of Oncological Diseases - Sofia District, Sofia
- Canada (9):
  - Cross Cancer Institute, Edmonton
  - qeii health sciences centre - VG site, Halifax
  - Juravinski Hospital and Cancer Centre, Hamilton
  - London Health Sciences Centre, London
  - Jewish General Hospital, Montreal
  - McGill University Health Centre, Montreal
  - R.S. McLaughlin Durham Regional Cancer Centre, Oshawa
  - Princess Margaret Cancer Centre, Toronto
  - British Columbia Cancer Agency-Vancouver Centre, Vancouver
- China (23):
  - Peking University First Hospital, Beijing
  - Chinese People's Liberation Army General Hospital - 301 Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - Chinese Academy of Medical Sciences Cancer Hospital, Beijing
  - 1st Hospital Jilin University, Changchun
  - Hunan Cancer Hospital - Xiangya Hospital - Central South University, Changsha
  - West China Hospital Sichuan University, Chengdu
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - The First Affiliated Hospital of Fujian Medical University, Fujian
  - Union Hospital of Fujian Medical University, Fuzhou
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - Zhejiang Provincial People's Hospital - Zhaohui, Hangzhou
  - Cancer Hospital of the University of Chinese Academy of Sciences Zhejiang Cancer Hospital, Hangzhou
  - Anhui Provincial Cancer Hospital, Hefei
  - Qilu Hospital of Shandong University, Jinan
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - Liaoning Cancer Hospital and Institute, Shenyang
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Affiliated Tumor Hospital of Xinjiang Medical University, Ürümqi
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
- Croatia (3):
  - Clinical Hospital Centre Split, Split
  - Clinical Hospital Centre "Sestre Milosrdnice", Zagreb
  - University Hospital Centre Zagreb, Zagreb
- Czechia (2):
  - Fakultni nemocnice Olomouc, Olomouc
  - Urocentrum Praha, Prague
- France (19):
  - Ramsay Health Clinic Belharra, Bayonne
  - CHU Saint Andre, Bordeaux
  - Centre Hospiltalier Universitaire Brest - Hôpital Morvan, Brest
  - Centre Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges- Francois Leclerc, Dijon
  - Centre Hospitalier Departemental Vendee, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Institut Régional du Cancer de Montpellier ICM Val d' Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Centre Hospitalier Universitaire de Nimes, Nîmes
  - Hôpital Européen Georges-Pompidou, Paris
  - Centre Eugene Marquis, Rennes
  - Centre Hospitalier Privé Saint-Grégoire, Saint-Grégoire
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Hôpital Foch, Suresnes
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Georgia (5):
  - High Technology Hospital MedCenter, Batumi
  - New Hospitals, Tbilisi
  - L. Managadze National Center of Urology, Tbilisi
  - Evex Medical corporation, Tbilisi
  - Jerarsi Clinic, Tbilisi
- Germany (10):
  - Universitatsklinik Dresden, Dresden
  - Malteser Waldkrankenhaus Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Centrum fur Hamatologie und Onkologie Bethanien, Frankfurt am Main
  - Asklepios Klinik Altona, Hamburg
  - Institut Für Versorgungsforschung in Der Onkologie, Koblenz
  - Universitatsklinikum Munster, Münster
  - Studienpraxis Urologie, Nürtingen
  - Universitätsklinikum Tübingen, Tübingen
  - Charité Universitätsmedizin Berlin - Campus Benjamin Franklin, Wien
- Greece (13):
  - 401 General Military Hospital of Athens, Athens
  - Henry Dunant Hospital, Athens
  - Alexandra General Hospital, Athens
  - Attikon Hospital, Chaïdári
  - Regional University General Hospital of Herakleio, Crete, Herakleio
  - University Hospital Of Ioannina, Ioannina
  - University Hospital of Larissa, Larissa
  - Athens Medical Center, Marousi
  - University Hospital of Patras, Pátrai
  - Bioclinic - Thessaloniki, Thessaloniki
  - Theagenio Anticancer Hospital of Thessaloniki, Thessaloniki
  - Anassa General Clinic, Thessaloniki
  - Interbalkan Medical Center of Thessaloniki, Thessaloniki
- Hong Kong (3):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Hong Kong United Oncology Centre, Kowloon
- Ireland (2):
  - Tallaght University Hospital, Dublin
  - University Hospital Waterford, Waterford
- Israel (7):
  - Shamir Medical Center (Assaf Harofeh), Be’er Ya‘aqov
  - Rambam Health Care Campus, Haifa
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Medical Center (Ichilov Hospital), Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (16):
  - Ospedale San Donato, Arezzo
  - Centro di Riferimento Oncologico di Aviano, Aviano
  - Istituto Tumori Bari Giovanni Paolo II - IRCCS, Bari
  - Istituto di Candiolo - Fondazione del Piemonte per l'Oncologia, Candiolo (TO)
  - Ospedale Policlinico San Martino, Genova
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliero Universitaria Maggiore Della Carita, Novara
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Istituto Regina Elena, Roma
  - Università Campus Bio-Medico di Roma, Rome
  - Ospedale Civile Di Sondrio, Sondrio
  - Azienda Ospedaliera Santa Maria di Terni, Terni
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Torino
  - Ospedale di Trento - Presidio Ospedaliero Santa Chiara, Trento
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Portugal (6):
  - Hospital de Braga, Braga
  - Unidade Local de Saúde da Guarda - Hospital Sousa Martins, Guarda
  - Centro Hospitalar de Leiria - Hospital de Santo André, Leiria
  - Centro Hospitalar de Lisboa Norte - Hospital de Santa Maria, Lisbon
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, E.P.E, Porto
  - Centro Hospitalar de Tras-os-Montes e Alto Douro, Vila Real
- BRCR Medical Center, Inc, San Juan, PR, Puerto Rico
- Singapore (3):
  - National University Hospital, Singapore
  - Icon Cancer Centre Farrer Park, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (13):
  - Pusan National University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Chungnam National University Hospital, Daejeon
  - National Cancer Center, Goyang-si
  - Pusan National University Yangsan Hospital, Gyeongsangnam-do
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul Saint Mary's Hospital, Seoul
  - The Catholic University of Korea Saint Vincent's Hospital, Suwon
- Spain (16):
  - Hospital del Mar - Parc de Salut, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Clínica Universidad de Navarra - Madrid, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda
  - Hospital Sant Joan de Déu de Manresa, Manresa
  - Complexo Hospitalario de Ourense (CHOU), Ourense
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville
  - Álvaro Cunqueiro Hospital, Vigo
- Sweden (3):
  - Länssjukhuset Ryhov, Jönköping
  - Universitetssjukhuset i Linköping, Linköping
  - Karolinska Universitetssjukhuset - Solna, Stockholm
- Switzerland (5):
  - University Hospital Basel, Basel
  - Istituto Oncologico Della Svizzera Italiana (IOSI), Bellinzona
  - University of Bern, Bern
  - Hôpitaux Universitaires de Genève, Geneva
  - Universitaetsspital Zurich - Klinik fur Medizinische Onkologie und Hematologie, Zurich
- Taiwan (10):
  - Chiayi Chang Gung Memorial Hospital, Buzi
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taipei Tzu Chi General Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou Branch, Taoyuan District
- Turkey (Türkiye) (8):
  - Hacettepe Universitesi Tip Fakultesi- Kanser Enstitusu, Ankara
  - Trakya Universitesi Saglik Arastirma ve Uygulama Merkezi, Edirne
  - Bagcilar Medipol Mega Universite Hastanesi, Istanbul
  - Istanbul Acibadem University Maslak Hospital, Istanbul
  - T.C. Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Medical Park Izmır Hastanesi, Izmir
  - Cebeci Hastanesi, Mamak
  - VKV Amerikan Hastanesi Department of Oncology, Şişli
- United Kingdom (13):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Dorset County Hospital NHS Foundation Trust, Dorchester
  - NHS Greater Glasgow and Clyde, Glasgow
  - Barts Health NHS Trust, London
  - Guys and Saint Thomas NHS Foundation Trust, Guy's Hospital, London
  - Sarah Cannon Research Institute London, London
  - The Christie NHS Foundation Trust, Manchester
  - East and North Hertfordshire NHS Trust, Middlesex
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Swansea Bay University Health Board, Port Talbot
  - Royal Preston Hospital, Preston
  - The Royal Marsden NHS Foundation Trust, Surrey
  - The Royal Wolverhampton NHS Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Powles T, Tagawa ST, Vulsteke C, Gross-Goupil M, Park SH, Necchi A, De Santis M, Duran I, Morales-Barrera R, Guo J, Sternberg CN, Bellmunt J, Goebell PJ, Kovalenko M, Boateng F, Sierecki M, Wang L, Sima CS, Waldes J, Bangs R, Loriot Y, Grivas P. A plain language summary of the TROPiCS-04 study: sacituzumab govitecan use after platinum-based chemotherapy and immunotherapy in people with locally advanced or metastatic cancer of the bladder, urethra, or upper urinary tract. Future Oncol. 2025 Dec;21(28):3593-3610. doi: 10.1080/14796694.2025.2579003. Epub 2025 Nov 23. PMID 41277126
- [Derived] Powles T, Tagawa S, Vulsteke C, Gross-Goupil M, Park SH, Necchi A, De Santis M, Duran I, Morales-Barrera R, Guo J, Sternberg CN, Bellmunt J, Goebell PJ, Kovalenko M, Boateng F, Sierecki M, Wang L, Sima CS, Waldes J, Loriot Y, Grivas P. Sacituzumab govitecan in advanced urothelial carcinoma: TROPiCS-04, a phase III randomized trial. Ann Oncol. 2025 May;36(5):561-571. doi: 10.1016/j.annonc.2025.01.011. Epub 2025 Feb 11. PMID 39934055
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=IMMU-132-13